CLINICAL TRIAL: NCT03814265
Title: Effect of Laughter Yoga on Mental Symptoms Frequency and Level of Saliva Cortisol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Fatma Ozlem Ozturk, Lecturer Fatma Ozlem Ozturk, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LYMSSC26102018
Record Dates: First submitted 2018-11-22; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Nursing Caries
Keywords: Cortisol; Laughter Yoga; Mental Symptom; Nursing; Student
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Laughter yoga group
  Interventions: Behavioral: Laughter yoga
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Laughter yoga — 440/5000 Laughter yoga; It is an exercise program that combines breathing techniques with unconditional laughter. During the sessions, laughter is simulated by hand clapping and warm-up exercises and by eye contact with other members in the group and by playing childish games with group members. Most of the time this simulation turns into genuine and contagious laughter. Laughter yoga is based on the argument that the brain cannot distinguish between real and unreal laugh.
  Arms: Intervention

SUMMARY:
The aim of this study is to evaluate the effect of laughter yoga on mental symptom frequency and salivary cortisol level among the 1st Year Nursing Students.

This is a randomized controlled study using pre-post-test design with control group. The population of our research; Ankara University Faculty of Health Sciences Nursing Department consisting of 202 students studying at the First Year.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of laughter yoga on mental symptom frequency and salivary cortisol level among the 1st Year Nursing Students.

This is a randomized controlled study using pre-post-test design with control group. The population of our research; Ankara University Faculty of Health Sciences Nursing Department consisting of 202 students studying at the First Year. A descriptive question form will apply to the entire population of the research.191 students fulfilling the criteria of this study will be included. Eleven students who have not fullfilled this criteria the inclusion criteria will be excluded from the study. Power analysis has been performed and the required sample volume for each group has been calculated as 34 with 0,90 power and 0.05 margin of error. Sample of the study consistsof 75 students considering the possibility of students leaving the research. This 75 students will be divided into two groups as intervention group (n=38) and control group (n=37). Intervention and control group have been randomly selected among Ankara University Faculty of Health Sciences Nursing Department.

ELIGIBILITY:
Inclusion Criteria:

* Ankara University Faculty of Health Sciences Department of Nursing to be a 1st year student.

Exclusion Criteria:

* Diabetes mellitus
* Hypertension
* Hypothyroidism
* Hyperaldosteronism
* Pregnancy
* Malignancy
* Congestive heart failure
* Psychotic disorder
* Chronic hepatic failure
* Nephrotic syndrome
* Chronic renal failure diagnosis
* Using medical drug

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Measurement of mental symptoms | Four weeks
  Data Collection Form is Brief Symptom Inventory(BSI). There are 5 sub-dimensions and 53 items in total.BSI has 5 sub-dimensions: Anxiety, Hostility, Somatization, Depression, Anxiety. The total score for each subscale is divided by the number of items in that sub-scale. The height of the total scores taken from the scale indicates the frequency of the individual's symptoms. The person answering the scale marks one of the following for each question: (0) None; (1) Very little; (2) "Moderate; (3) quite a lot; (4) Too much Application process consist of three phases such as; pre-test, intervention and post-test. During pre-test phase. Whether there is a significant decrease in posttest scores compared to pre-test mean scores.

SECONDARY OUTCOMES:
Measurement of saliva cortisol | Each session for four weeks
  Saliva samples for the study of salivary cortisol level. Saliva samples have been taken from intervention and control group students for measurement of salivary cortisol level at 07.55 am before each session. During the intervention phase; laughter yoga has been applied to the intervention group after the pre-test. There hasn't been any intervention for the control group during the research.Saliva samples have been taken from the students who have participated in the study at 08.40 am for each cortisol level measurement after each session. According to the Preliminary Test, it will be evaluated whether there is a significant decrease in the final test scores.

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer Tezel, Prof. Dr., Study Director — Ankara Uviversity
Locations (1):
- Ankara University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT03814265/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT03814265/SAP_001.pdf
  • Informed Consent Form (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT03814265/ICF_002.pdf